CLINICAL TRIAL: NCT03256903
Title: Open Randomized Clinical Trial to Compare Pain Relief Between Methoxyflurane and Standard of Care for Treating Patients With Trauma Pain in Spanish Emergency Units.
Brief Title: Methoxyflurane vs Standard Analgesic Treatment for Trauma Pain in Spanish Emergency Units
Acronym: InMEDIATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Pharmaceuticals S.L. (Industry)
Collaborators: Spanish Society for Emergency Medicine (SEMES) (Unknown); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Principal Investigator, Alberto M. Borobia, MD, PhD, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR311-3502
Record Dates: First submitted 2017-05-30; First posted 2017-08-22 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Acute Pain Due to Trauma
Keywords: Methoxyflurane; emergency; trauma pain; inhaled analgesia
MeSH Terms: conditions — Emergencies | interventions — Methoxyflurane; Standard of Care

STUDY DESIGN:
Intervention Model Description: Phase IIIb open randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methoxyflurane (Experimental): Patients will be supplied with up to two inhalers containing 3 mL methoxyflurane. A member of the research team will train the patient to self-administer methoxyflurane
  Interventions: Drug: Methoxyflurane
- Standard of Care (SoC) (Active Comparator): Patients will be treated following standard of care (SoC) of the hospital, for emergency relief of trauma and associated pain. Any kind of analgesia administered by any route will be valid. Only administration of one analgesic (or fixed combinations) at baseline will considered SoC. Other required analgesics will be considered rescue medication.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Methoxyflurane — Up to two inhalers containing 3 mL methoxyflurane. Treatment duration: 1 administration in 1 day.
  Other Names: No other interventions
  Arms: Methoxyflurane
Drug: Standard of care — Any kind of analgesia, administered by any route for emergency relief of moderate to severe pain in conscious adult patients with trauma and associated pain
  Other Names: No other interventions
  Arms: Standard of Care (SoC)

SUMMARY:
Clinical trial to compare pain relief between methoxyflurane and any analgesic treatment used in usual clinical practice, in patients with trauma and associated pain, treated in Spanish emergency units.

DETAILED DESCRIPTION:
Open, randomized clinical trial to compare emergency pain relief between methoxyflurane and standard of care in patients with trauma and associated pain, treated in Spanish emergency units.

Methoxyflurane is a fluorinated ethyl methyl ether, with the chemical name 2:2-dichloro-1:1-difluoroethyl methyl ether. It belongs to the fluorinated hydrocarbon group of volatile anaesthetics. It is inhaled as a vapour at low (sub-anaesthetic) concentrations to achieve an analgesic effect for the management of pain.

In Europe countries, where methoxyflurane is already marketed, it is indicated for emergency relief of moderate to severe pain in conscious adult patients with trauma and associated pain.

On the other hand, current clinical practice includes a variety of analgesic agents, with the choice of which to employ based on consideration of the risk-benefit factors of each class of drug, as well as the type of pain, its severity, and the risk of adverse effects.

The main objective of this study is to assess Methoxyflurane's significant advantage in terms of anaglesic effectiveness, as it is known as a rapidly acting, non-narcotic analgesic for the treatment of emergency pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients: ≥ 18 years of age
* Moderate to severe pain (NRS 0-10; >=4) secondary to trauma
* Without anticipating surgery due to the trauma, requiring hospitalization (hospital stay 12h)
* Conscious patient.
* Giving informed consent in writing

Exclusion Criteria:

* Hypersensitivity to methoxyflurane (MEOF) or any fluorinated anaesthetic.
* Malignant hyperthermia: patients with known or genetically susceptible to malignant hyperthermia or a history of severe adverse reactions in either patient or relatives.
* Patients who have a history of showing signs of liver damage after previous MEOF use or halogenated hydrocarbon anaesthesia
* Known clinically significant renal impairment
* Known pregnant or likely to be pregnant women at the time of inclusion.
* Clinically evident cardiovascular instability
* Clinically evident respiratory depression
* Patients taken any analgesic for the traumatic pain before inclusion
* Altered level of consciousness due to any cause, including head injury, drugs or alcohol
* Degenerative diseases, mental illness or other conditions that could affect ability of valuing pain intensity
* Patients to be unable to understand the purpose of the study and perform self-assessments, following investigator's criteria.
* Participation in another clinical trial within 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Pain relief | At baseline, 3, 5, 10, 15 and 20 minutes from STA
  Change in mean pain intensity over 20 min from start of administration (STA) and time to first pain relief, measured by numeric scale (0-10)
Analgesia effectiveness | Change from baseline to 3, 5, 10, 15, 20 and 30 min
  Difference between arms related to analgesia effectiveness
Analgesia speed of action | From time of randomization up to 20 minutes
  Difference between arms related to speed of action of analgesia for all patients
Safety for patients with severe pain, treated with second or third step analgesics | Up until 14 days from STA
  Difference between arms related to safety for patients with severe pain (NRS >7), treated with second or third step analgesics
Patient-averaged summed pain intensity difference 15 min after STA | from baseline to 3, 5, 10 and 15 minutes post dose
  Patient-averaged summed pain intensity difference 15 min after STA
Pain Responders | from baseline to 20 minutes post dose
  Pain Responders (with >30% pain relief compared to baseline) at 20 min

SECONDARY OUTCOMES:
Investigators and patients satisfaction | 30 min from start of administration
  Investigators and patients satisfaction measured as convenience, treatment efficacy and adverse events, using NRS scales (0-10)
Patient and investigators' fulfillment of expectations | 30 min from start of administration
  Patient and investigators' fulfillment of expectations, measured with a 5 items Likert scale
Patients' Global Impression of Change with the treatments | Up until 30 minutes from STA
  Patients' Global Impression of Change with the treatments, measured using a 7 items Likert scale
Treatment cost of pain relief | Up until 60 minutes from randomization
  Treatment cost of pain relief, measured considering use of fungible material; need of nurse to administer iv treatments; time to discharge
Safety rates of treatment emergent adverse events | Up until 14 days from STA
  Safety rates of treatment emergent adverse events (TEAE) in both arms, including alterations in biochemical and blood count.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Borobia, MD, PhD, Study Director — La Paz University Hospital
Locations (14):
- Spain (14):
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital del Bierzo, Ponferrada, León
  - Hospital Asepeyo Coslada, Coslada, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Gernika-Lumo, Gernika-Lumo, Vizcaya
  - Hospital General de Alicante, Alicante
  - Hospital Universitario La Princesa, Madrid
  - Hospital Clínico San Carlos, Madrid
  - SUMMA - Comunidad de Madrid, Madrid
  - Hospital La Paz, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital Campo Grande, Valladolid
  - Complejo Asistencial de Zamora, Zamora

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Borobia AM, Collado SG, Cardona CC, Pueyo RC, Alonso CF, Torres IP, Gonzalez MC, Casal Codesido JR, Betegon MA, Barcela LA, Andicoechea AO, Testa AF, Colina JT, Dorribo AC, Del Arco Galan C, Martinez Avila JC, Lugilde ST, Carcas Sansuan AJ; InMEDIATE Investigators Group. Inhaled Methoxyflurane Provides Greater Analgesia and Faster Onset of Action Versus Standard Analgesia in Patients With Trauma Pain: InMEDIATE: A Randomized Controlled Trial in Emergency Departments. Ann Emerg Med. 2020 Mar;75(3):315-328. doi: 10.1016/j.annemergmed.2019.07.028. Epub 2019 Oct 14. PMID 31623936